CLINICAL TRIAL: NCT03021434
Title: Cluster Randomized Trial of Low-cost Microbiological Water Test Kits
Brief Title: Trial of Low-cost Microbiological Water Test Kits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Indian Institute of Technology Kanpur (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11920/RR/5743
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-01

CONDITIONS: Diarrhea; E.Coli Infections
Keywords: Water Supply/standards; Water microbiology; India; Hand disinfection; Escherichia coli Infections/prevention & control; Hygiene; Health behavior; Drinking water; Informational intervention
MeSH Terms: conditions — Diarrhea; Escherichia coli Infections; Health Behavior | interventions — Residence Characteristics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard Testing (Experimental): Households will participate in community and household water safety education sessions, during which they will be given generalized information on water quality and safe water handling. A water sample from these households will be collected for laboratory analysis. Household-specific water quality information will be delivered to households within 72 hours, and households will be informed whether their drinking water was found to be contaminated. A study team member will review the information from the laboratory tests with the household and review information covered in the informational materials on safe water handling, storage, and use behaviours.
  Interventions: Other: Community and household water safety education sessions; Other: Household-specific water quality information
- Test Kits (Experimental): Households will participate in community and household water safety education sessions, during which they will be given generalized information on water quality and safe water handling. Data collectors will demonstrate the use of the low-cost microbiological water test kits and test household stored drinking water. A study team member will return to the household within 72 hours and review the household-specific water quality information from the initial test with household members. Households will be given 10 water test kits to use at their discretion over the 1-2 month follow up period. They will be appropriately trained in how to both perform the test and interpret the results. Households will also review information on safe water handling, storage, and use behaviours.
  Interventions: Other: Community and household water safety education sessions; Other: Household-specific water quality information; Other: Low-cost microbiological water test kits
- Comparison (Active Comparator): Households will participate in community and household water safety education sessions, during which they will be given generalized information on water quality and safe water handling. A water sample from these households will be collected for laboratory analysis. Results from this analysis will be returned to the household at project endline. A study team member will return to the household within 72 hours to review the information on safe water handling, storage, and use behaviours.
  Interventions: Other: Community and household water safety education sessions

INTERVENTIONS:
Other: Community and household water safety education sessions — Data collectors will give a short community presentation on water treatment, as well as safe water handling and storage. Then, data collectors will immediately visit households and review this information. Data collectors will return within 72 hours and review this information once more.
Other: Household-specific water quality information — Household specific water quality data will be provided in two ways. In the Standard Testing Arm, water quality data will be analyzed in a laboratory by standard methods and results will be delivered to households. In the Test Kit arm, water quality data will be analyzed in households using provided water test kits.
  Arms: Standard Testing; Test Kits
Other: Low-cost microbiological water test kits — Intervention component consists of low-cost, biodegradable that tests for the presence of E. coli in water samples. The test uses Aquatest broth medium with resorufin methyl ester chromogen. Presence of E. coli (positive test) imparts bright red color, making it easy to use/interpret at the household level with minimal training
  Arms: Test Kits

SUMMARY:
The present study is a cluster randomized control trial of low-cost microbiological water test kits in rural and peri-urban communities in the Kanpur region of Uttar Pradesh, India.

DETAILED DESCRIPTION:
The proposed trial utilizes a cluster randomized controlled methodology, with clustering occurring at the village level. The intervention that will be tested in this cluster randomized controlled trial is informed by the development of a simple, low-cost water quality test kit developed and piloted by J. Brown and colleagues in Nagpur, Maharashtra.

There will be two intervention arms and one control/comparison arm. In all selected villages, the study team will work with local government to conduct a village-level information session on water quality and key water safety behaviours. Informational material on water safety behaviours will be distrubted to all houseohlds following this information session. In the control group, households will be visited to provide water safety informational cards and collect a drinking water sample to be analyzed in the lab. They will not receive the results of the analysis until the conclusion of the study. Households in Intervention Arm 1 (Standard Testing) will have their water sampled and analyzed in the lab, and results of the analysis will be delivered to the households. They will receive informational cards describing water purification strategies. Households in Intervention Arm 2 (Test Kits) will be provided with the materials and training needed to perform water quality testing in their own household using the newly developed testing kits. They will also receive informational cards describing water purification strategies.

Following the initial village-level information session, the study team will randomly sample households for participation in the trial. Participating households will complete a short survey on household demographics and water handling, storage, and use behaviours and a water sample will be taken and tested in the lab for fecal indicator bacteria. At an unannounced follow-up visit, roughly 1 - 2 months after enrollment, households will complete a short survey about changes in water handling, storage, and use behaviours and a second sample of household stored drinking water will be collected for laboratory analysis. The effect of the cluster randomized controlled trial on water quality will be determined by comparing arithmetic mean E. coli count from samples of household water and changes in water safety behaviours between baseline and endline.

Microbiological drinking water quality will be assessed at two time points: baseline and endline. At each visit, a 330 ml sample of household water will be collected for analysis; we will ask participants to fill the sample container as if it were a drinking cup for a child living in the household. Samples will be kept cold (on ice in a cooler) until delivery to the laboratory and thereafter stored at 4oC until processing, to begin within 8 hours of the sampling event.

ELIGIBILITY:
Inclusion Criteria (for villages) :

* Village located within the Kanpur district, within
* Village population between 100 and 1000 households.
* No chlorinated water sources available in the village.

Inclusion Criteria (for households) :

* Consent to participate in the study
* Contain at least one child who is between 29 days and 60 months of age at the time of enrollment

Exclusion Criteria:

* Villages that receive chlorinated water from utility services

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 572 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05-25 (Actual); Study Completion 2017-05-25 (Actual)

PRIMARY OUTCOMES:
Arithmetic mean E. coli count from sample of stored household drinking water | 1-2 month follow up visit post initial household information session
  A sample of household drinking water will be collected and analyzed in a standard laboratory using membrane filtration.

SECONDARY OUTCOMES:
Water storage, handling, and use behaviors | 1-2 month follow up visit post initial household information session
  Self-reported water treatment practices, verifiable water treatment practices, water handling and water storage practices in the home, and changes in primary water source. This outcome is measured using baseline and follow up survey questionnaires, as well as direct observation of handwashing station and water storage containers
Intervention uptake/use | 1-2 month follow up visit post initial household information session
  For households participating in the Test Kit Arm, intervention update will be assessed visual inspection of the number of test kits remaining in the household at end line (to determine utilization) as well as targeted survey question on the ease of use and perceived utility of the test kits.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Dreibelbis, PhD, Principal Investigator — London School of Hygiene and Tropical Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kotloff KL, Nataro JP, Blackwelder WC, Nasrin D, Farag TH, Panchalingam S, Wu Y, Sow SO, Sur D, Breiman RF, Faruque AS, Zaidi AK, Saha D, Alonso PL, Tamboura B, Sanogo D, Onwuchekwa U, Manna B, Ramamurthy T, Kanungo S, Ochieng JB, Omore R, Oundo JO, Hossain A, Das SK, Ahmed S, Qureshi S, Quadri F, Adegbola RA, Antonio M, Hossain MJ, Akinsola A, Mandomando I, Nhampossa T, Acacio S, Biswas K, O'Reilly CE, Mintz ED, Berkeley LY, Muhsen K, Sommerfelt H, Robins-Browne RM, Levine MM. Burden and aetiology of diarrhoeal disease in infants and young children in developing countries (the Global Enteric Multicenter Study, GEMS): a prospective, case-control study. Lancet. 2013 Jul 20;382(9888):209-22. doi: 10.1016/S0140-6736(13)60844-2. Epub 2013 May 14. PMID 23680352
- [Background] Million Death Study Collaborators; Bassani DG, Kumar R, Awasthi S, Morris SK, Paul VK, Shet A, Ram U, Gaffey MF, Black RE, Jha P. Causes of neonatal and child mortality in India: a nationally representative mortality survey. Lancet. 2010 Nov 27;376(9755):1853-60. doi: 10.1016/S0140-6736(10)61461-4. Epub 2010 Nov 12. PMID 21075444
- [Background] Lakshminarayanan S, Jayalakshmy R. Diarrheal diseases among children in India: Current scenario and future perspectives. J Nat Sci Biol Med. 2015 Jan-Jun;6(1):24-8. doi: 10.4103/0976-9668.149073. PMID 25810630
- [Background] Hamoudi A, Jeuland M, Lombardo S, Patil S, Pattanayak SK, Rai S. The effect of water quality testing on household behavior: evidence from an experiment in rural India. Am J Trop Med Hyg. 2012 Jul;87(1):18-22. doi: 10.4269/ajtmh.2012.12-0051. PMID 22764286
- [Background] Davis J, Pickering AJ, Rogers K, Mamuya S, Boehm AB. The effects of informational interventions on household water management, hygiene behaviors, stored drinking water quality, and hand contamination in peri-urban Tanzania. Am J Trop Med Hyg. 2011 Feb;84(2):184-91. doi: 10.4269/ajtmh.2011.10-0126. PMID 21292883
- [Background] Dufour AP, Strickland ER, Cabelli VJ. Membrane filter method for enumerating Escherichia coli. Appl Environ Microbiol. 1981 May;41(5):1152-8. doi: 10.1128/aem.41.5.1152-1158.1981. PMID 7020592
- [Background] Brown J, Stauber C, Murphy JL, Khan A, Mu T, Elliott M, Sobsey MD. Ambient-temperature incubation for the field detection of Escherichia coli in drinking water. J Appl Microbiol. 2011 Apr;110(4):915-23. doi: 10.1111/j.1365-2672.2011.04940.x. PMID 21214694
- [Background] Bain RE, Woodall C, Elliott J, Arnold BF, Tung R, Morley R, du Preez M, Bartram JK, Davis AP, Gundry SW, Pedley S. Evaluation of an Inexpensive Growth Medium for Direct Detection of Escherichia coli in Temperate and Sub-Tropical Waters. PLoS One. 2015 Oct 23;10(10):e0140997. doi: 10.1371/journal.pone.0140997. eCollection 2015. PMID 26495983
- [Background] Magro G, Bain RE, Woodall CA, Matthews RL, Gundry SW, Davis AP. Synthesis and application of resorufin beta-D-glucuronide, a low-cost chromogenic substrate for detecting Escherichia coli in drinking water. Environ Sci Technol. 2014 Aug 19;48(16):9624-31. doi: 10.1021/es502319n. Epub 2014 Jul 29. PMID 25035967
- [Background] Creswell, J.W. and V.L. Plano Clark, Designing and conducting mixed methods research. 2011, Los Angeles: SAGE Publications.
- [Background] Haas, C.N., How to average microbial densities to characterize risk. Water Research, 1996. 30(4): p. 1036-1038.
- [Background] Moher D, Schulz KF, Altman DG; CONSORT Group (Consolidated Standards of Reporting Trials). The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomized trials. J Am Podiatr Med Assoc. 2001 Sep;91(8):437-42. doi: 10.7547/87507315-91-8-437. PMID 11574648
- [Background] Witte, K., Putting the fear back into fear appeals: The extended parallel process model. Communications Monographs, 1992. 59(4): p. 319-26.
- [Background] Hayes RJ, Bennett S. Simple sample size calculation for cluster-randomized trials. Int J Epidemiol. 1999 Apr;28(2):319-26. doi: 10.1093/ije/28.2.319. PMID 10342698
- [Background] Duflo, E., R. Glennerster, and M. Kremer, Using Randomization in Development Economics Research: A Toolkit, in T. Schultz and John Strauss, eds., Handbook of Development Economics. 2008, North Holland: Amsterdam and New York.
- [Background] Fleiss, J.L., Appendix: Sample-Size Determination, in The Design and Analysis of Clinical Experiments. 1999, John Wiley & Sons, Inc. p. 369-417.
- [Background] Zhou H, Taber C, Arcona S, Li Y. Difference-in-Differences Method in Comparative Effectiveness Research: Utility with Unbalanced Groups. Appl Health Econ Health Policy. 2016 Aug;14(4):419-429. doi: 10.1007/s40258-016-0249-y. PMID 27371369
- [Background] Graneheim UH, Lundman B. Qualitative content analysis in nursing research: concepts, procedures and measures to achieve trustworthiness. Nurse Educ Today. 2004 Feb;24(2):105-12. doi: 10.1016/j.nedt.2003.10.001. PMID 14769454
- [Background] Burnard P. A method of analysing interview transcripts in qualitative research. Nurse Educ Today. 1991 Dec;11(6):461-6. doi: 10.1016/0260-6917(91)90009-y. PMID 1775125